CLINICAL TRIAL: NCT04796506
Title: Slow Wave Sleep As a Biomarker of Rehabilitation-induced Cognitive Improvement in Parkinson's Disease R01 HD100670
Brief Title: Slow Wave Sleep As a Biomarker of Rehabilitation-induced Cognitive Improvement in PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 22-1685; IRB-300005901 (Other: UAB IRB); R01HD100670 (NIH)
Record Dates: First submitted 2020-11-30; First posted 2021-03-15 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: PD subjects will be randomized (1:1) to the progressive resistance training (PRT) rehabilitation group or the delayed exercise (DE) control group (wait 12 weeks and begin resistance training). Change in slow wave sleep (SWS) from baseline to 12-weeks will be used to determine the arm assignment in the second 12-week period of the trial for the original PRT group. Specifically, participants with an increase in SWS (responders) will continue in PRT for the 2nd 12 weeks of the trial, while non-responders (participants without increase in SWS) will transition to endurance training (ET) to assess if PRT followed by ET can enhance response in these non-responders.
Who Masked: Outcomes Assessor
Masking Description: Interpretation of polysomnography and cognitive performance will be blinded to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (Active Comparator): PD participants randomized to progressive resistance training PRT) will have 12 weeks of supervised PRT 3 times per week. After the 1st 12 weeks, responders to PRT (increase in slow wave sleep) will continue PRT for an additional 12 weeks, non-responders to PRT will transition to endurance training (ET).
  Interventions: Other: Progressive Resistance Training (PRT); Other: Endurance Training (ET)
- Delayed Exercise Group (Placebo Comparator): PD participants randomized to the delayed exercise control group will not exercise for the 1st 12 weeks of the study. After the 1st 12 weeks, participants in the delayed exercise group will transition to PRT for the 2nd 12 weeks.
  Interventions: Other: Progressive Resistance Training (PRT); Other: Delayed Exercise Training (DE)

INTERVENTIONS:
Other: Progressive Resistance Training (PRT) — PD subjects may be randomized (1:1) to PRT with supervised sessions 3 times per week for 12 weeks. Exercise training will consist of a combination of resistance training (RT) and bodyweight functional mobility exercises with limited rest intervals. The full volume exercise prescription will consist of: 1) five movements to improve strength and muscle mass each performed for 3 sets of 8-12 repetitions; 2) trunk exercises to improve postural stability; and 3) 3-4 bodyweight exercises to improve power and balance. Change in slow wave sleep (SWS) from baseline to 12-weeks will be used to determine the assignment in the second 12-week period. Subjects with an increase in SWS by >24 minutes will continue in PRT for the 2nd 12 weeks of the trial, while participants with <24 minutes increase in SWS will transition to endurance training (ET).
  Other Names: PRT
Other: Delayed Exercise Training (DE) — PD subjects randomized to the exercise control group (1:1) will not exercise during the first 12 weeks of the study. During that time, they will be asked not to change their physical activity levels or dietary habits. All participants in the delayed-exercise group will begin PRT at completion of the 1st 12-week period.
  Arms: Delayed Exercise Group
Other: Endurance Training (ET) — Non-responders to PRT will transition too ET during 2nd 12 weeks of the study. This intervention is supervised endurance training, 3 times per week for 12 weeks. Each session lasts approximately 75 min., comprised of warm-up, stimulus phase for 50-60 min., and cool-down. Sessions are split between cycle ergometer and treadmill exercise. Participant heart rate is monitored to maintain target exercise intensity of 60-80% (±5%) of heart rate reserve (HRR).
  Other Names: ET
  Arms: Exercise Group

SUMMARY:
The purpose of this study is to investigate the effects of exercise rehabilitation on cognition and to evaluate slow wave sleep (SWS) as a biomarker and mediator of response to rehabilitation-induced improvement in cognitive performance among persons with Parkinson's disease (PwP), with the ultimate goal of maximizing rehabilitation efficacy at the individual level (i.e. precision rehabilitation).

DETAILED DESCRIPTION:
Sleep impairment adversely affects cognitive function and increases risk for dementia. Slow wave sleep (SWS) or delta sleep (non-rapid eye movement (REM) stage 3; N3) is especially important for cognition due to its association with synaptic plasticity, synaptic potentiation, synaptic renormalization, and cortical reorganization, especially in prefrontal cortex. Clinically, SWS contributes to memory consolidation and language performance. The investigators have previously shown that the amount of SWS in persons with Parkinson's disease (PwP) is related to cognitive performance, especially in the domain of executive function. The investigators have also shown that exercise increases SWS in some PwP and that participants who have an exercise-induced increase in SWS also have improvement in executive function. This study will evaluate changes in cognitive function and SWS due to progressive resistance training rehabilitation (PRT). Participants who do not have an increase in SWS with PRT (non-responders) over 12 weeks will be transitioned to an endurance training (ET) intervention, while those who do have an increase in SWS (responders) will continue in PRT for an additional 12 weeks.

ELIGIBILITY:
Inclusion:

* clinical diagnosis of idiopathic PD, based on the presence of bradykinesia as well as at least one of the following: rest tremor, rigidity, and/or postural instability (per United Kingdom PD Brain Bank Criteria)
* Hoehn and Yahr stage 2-3 (performed at screening visit)
* age ≥ 45 and
* on stable medications for at least 4 weeks prior to study entry without expecting to change medications for the duration of the study.
* Montreal Cognitive Assessment (MoCA) score ≥ 18 and <26 (performed at screening visit)
* No contraindications to an exercise program.

Exclusion:

* fails exercise readiness evaluation at screening visit
* regular participation in an exercise program
* cardiovascular or pulmonary disease, including uncontrolled hypertension, congestive heart failure, unstable coronary artery disease, serious arrhythmia, stroke within the past year, or chronic obstructive pulmonary disease (COPD)
* shift workers
* signs indicative of atypical Parkinsonism (cerebellar signs, supranuclear gaze palsy, apraxia, prominent autonomic failure, or other cortical signs)
* secondary Parkinsonism (neuroleptic treatment at time of onset of Parkinsonism or at time of study entry, history of multiple strokes with stepwise progression of Parkinsonism, or history of multiple head injuries)
* inability to walk without assistance
* deep brain stimulation (DBS)
* known narcolepsy
* untreated sleep apnea
* any condition that, in the opinion of the investigator, will preclude the participant from successfully or safely completing study procedures.

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition in Stroop inhibition | Baseline to twelve weeks
  Change in executive function on the Stroop inhibition

SECONDARY OUTCOMES:
Change in slow wave sleep (SWS) | Change from baseline to twelve week and change from twelve weeks to 24 weeks.
  Change in slow wave sleep as measured by polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Amy Amara, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No